CLINICAL TRIAL: NCT03806309
Title: A Randomized Non-comparative Phase II Study of Maintenance Therapy With OSE2101 Plus FOLFIRI, or FOLFIRI After Induction Therapy With FOLFIRINOX in Patients With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma (TEDOPaM-D17-01 PRODIGE 63 Study)
Brief Title: OSE2101+FOLFIRI, or FOLFIRI Maintenance After FOLFIRINOX-based Induction Therapy in Advanced or Metastatic PDAC
Acronym: TEDOPAM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: OSE Immunotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEDOPAM D17-01 PRODIGE 63
Record Dates: First submitted 2018-11-24; First posted 2019-01-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Locally Advanced Cancer; Metastatic Cancer
Keywords: Immunotherapy; Chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — IFL protocol; Leucovorin; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : maintenance with FOLFIRI (Active Comparator): FOLFIRI (IV; folinic acid 400 mg/m^2, irinotecan 180 mg/m^2, 5-FU bolus 400 mg/m^2 and continuous infusion 2,400 mg/m^2/46h (dose adjustment will be accepted).
  Interventions: Drug: FOLFIRI
- Arm B : maintenance with OSE2101 plus FOLFIRI (Experimental): OSE2101 - subcutaneous injection on day 1 and day 15, every 4 weeks for 6 doses then every 8 weeks until month 12 then every 12 weeks up to 24 months.
  FOLFIRI - schedules as in Arm A until disease progression on unacceptable toxicity
  Interventions: Drug: FOLFIRI; Drug: OSE2101

INTERVENTIONS:
Drug: FOLFIRI — Intravenous (IV); folinic acid 400 mg/m^2, irinotecan 180 mg/m^2, 5-FU bolus 400 mg/m^2 and continuous infusion 2,400 mg/m^2
  Other Names: Leucovorin (Folinic Acid), Fluorouracil, Irinotecan
Drug: OSE2101 — subcutaneous injection on days 1 and 15, every 4 weeks for 6 doses then every 8 weeks until month 12 and then every 12 weeks for a maximum treatment duration of 24 months
  Other Names: Tedopi
  Arms: Arm B : maintenance with OSE2101 plus FOLFIRI

SUMMARY:
TEDOPAM is a randomized (1.1.1) non-comparative phase II study. This study will assess the efficacy and safety of OSE2101 alone or in combination with nivolumab followed by FOLFIRI reintroduction, versus FOLFIRI as maintenance therapy in patients with advanced PDAC after induction therapy with FOLFIRINOX.

DETAILED DESCRIPTION:
Current standard of care for patients with advanced pancreatic ductal adenocarcinoma (PDAC) is chemotherapy, preferential regimen being FOLFIRINOX (5FU, leucovorin, irinotecan, and oxaliplatin) in fit patients (PS 0-1, bilirubin < 1.5 ULN). The question of how and when the FOLFIRINOX regimen and doses can be deescalated after a period of disease control (i.e. maintenance therapy) remains unanswered. In routine practice, oxaliplatin is usually stopped after 6-8 cycles due to limiting neuropathy, and the fluoropyrimidine is continued, either alone or, more frequently, in combination with irinotecan (FOLFIRI regimen), until disease progression.

Immune therapies have opened new opportunities in cancer therapy. However, results of immunotherapy in PDAC have been disappointing so far, with failure of checkpoint inhibitor monotherapies (anti-CTLA4 and anti-PD-L1 monoclonal antibodies [mAb]) in progressive advanced PDAC, while monovalent vaccines were demonstrated to be safe but with limited activity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent document, willing and able to comply with protocol requirements,
2. Histologically or cytologically proven pancreatic ductal adenocarcinoma,
3. Age ≥ 18 years,
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1,
5. Human Leukocyte Antigen (HLA-A2) genotype,
6. Recurrent or advanced disease not amenable to surgery with curative intent (previous resection of primary tumor allowed),
7. Measurable or evaluable (radiologically detectable disease which does not fulfill RECIST criteria for measurable disease) lesions according to RECIST v1.1 criteria (CT-scan < 4 weeks),
8. Stable disease or tumor response according to RECIST v1.1 after a 4-month (8 cycles) course of first-line FOLFIRINOX or modified FOLFIRINOX induction chemotherapy,
9. Have archival tissue sample that has been identified and confirmed as available for study, or newly obtained core or excisional biopsy of a tumor lesion,
10. Adequate organ function, as defined by the following:

    * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN),
    * Total serum bilirubin < 1.5 ULN,
    * Prothrombin ratio > 70%,
    * Serum albumin ≥ 2.8 g/dL,
    * Hemoglobin ≥ 10,0 g/dl,
    * White blood cell count (WBC) ≥ 3,000/μL,
    * Absolute neutrophil count (ANC) ≥ 1,500/μL,
    * Platelets ≥ 100,000/μL,
    * Serum creatinine ≤ 1.5 ULN or creatinine clearance > 50 mL/min (Modification of diet in renal disease [MDRD]),
11. Life expectancy ≥ 3 months,
12. Women participants of childbearing potential must have a negative serum pregnancy test within the 3 days prior to the first treatment administration. Both women participants of childbearing potential and men participants who are sexually active with women of childbearing potential must agree to use a reliable method of birth control (i.e. pregnancy rate < 1% per year) until 6 months after the last dose of FOLFIRI, and 90 days after the last dose of OSE2101,
13. Registration in a national health care system (PUMA included).

Exclusion Criteria:

1. Obstructive jaundice (bilirubin > 1.5 ULN) without adequate biliary drainage,
2. Allograft recipient,
3. Active HBV (hepatitis B virus), HCV (hepatitis C virus ), or HIV infection, Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive HBc (hepatitis B core antigen) antibody test are eligible.

   Note: Patients positive for HCV antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA).
4. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri,
5. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of neuropathy, alopecia, and the laboratory values defined in the inclusion criteria,
6. Known active central nervous system metastases and/or carcinomatous meningitis; patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurological symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids at a dose > 10 mg/day of prednisone or equivalent for at least 14 days prior to trial treatment,
7. Uncontrolled massive pleural effusion or massive ascites,
8. Evidence of interstitial lung disease, any active, non-infectious pneumonitis, or known active tuberculosis,
9. Active uncontrolled infection, or current unstable or uncompensated respiratory or cardiac conditions, or bleeding,
10. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study,
11. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant, in the opinion of the treating investigator,
12. Known or suspected drug hypersensitivity to OSE2101 vaccine,
13. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug,
14. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational product, Note: Local surgery of isolated lesions for palliative intent is acceptable.
15. Treatment with any investigational medicinal product within 28 days prior to study entry,
16. Prior intolerance/severe toxicity with 5-fluorouracil (5-FU) or irinotecan (including dihydropyrimidinedehydrogenase [DPD] and UGT1A1 deficiency),
17. Pregnancy/lactation,
18. Tutelage or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | At 12 months
  The OS is defined according to the DATECAN (Definition for the Assessment of Time-to-event Endpoints in CANcer trials) consensus as the time from randomization to death for any reason. In the absence of confirmation of death, survival time will be censored at the date of the last clinical assessment

SECONDARY OUTCOMES:
Progression free survival (PFS) by centralized review of CT-scan imaging. | assessed up to 60 months
  The PFS is defined according to the DATECAN consensus as the time from randomization to first progression or death for any reason, whichever occurs first. In the absence of event (confirmation of progression or death), PFS status will be censored at the date of the last radiological assessment.
  PFS according to RECIST (Response Evaluation Criteria In Solid Tumors) v1.1 in the FOLFIRI arm (Arm A) and iRECIST (immune Response Evaluation Criteria In Solid Tumors) in the immune therapy arms (Arm B and C) by centralized review of CT-scan imaging
Rate of patients with success of the strategy (SSR) | At 6 months
  The SSR is derived from the duration of disease control (DDC), which is defined as the PFS, or, if FOLFIRI is reintroduced and achieves partial response (PR) or stable disease (SD), as the addition of the initial PFS (PFS1) and the PFS of the reintroduction PFS (PFS2)
Number of participants with treatment-related adverse events as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events [NCICTCAE] v5.0 | from signature of informed consent to 28 days after the last administration of the investigational product in Arm A and B and 100 days after the last administration of the investigational product in Arm C.
  All grade and severe (grade 3-5) toxicities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Objective response rate (ORR) | assessed up to 60 months
  Response according to RECIST v1.1 in the FOLFIRI arm (Arm A) and iRECIST in the immune therapy arms (Arms B and C) (centralized review of CT-scan imaging); a comparative analysis of tumor response according to these two evaluation rules will be performed in Arm B and C
Health-related Quality of life (HRQoL) evaluation assessed by EORTC QLQ (quality of life questionnaire) -C30 questionnaire | Baseline, Month 2, Month 4, Month 6, Month 8, Month 10, Month 12, Month 14, Month 16, Month 18, Month 20, Month 22, Month 24 (until the date of first documented progression or date of death, assessed up 60 months)
  Rate of patients with an improvement of their quality of life score according to EORTC QLQ-C30. A quality of life score is obtained according to the answers to the 30 questions. The Minimal Clinically Important Difference (MCID) will be fixed to 10 points.
Estimate the Quality-Adjusted Time Without Symptoms of Disease or Toxicity of Treatment (Q-Twist) for each participant | assessed up to 60 months
  Q-TWiST analysis considers three health states, TOX (toxicity), TWiST, and REL (The duration of the relapse), and the duration of each state is calculated for every patient.
  The TOX state comprises the total number of days after randomisation and before strategy failure spent with toxicity, regardless of when the toxicity started or whether there were gaps between toxicities. All grade 3 or 4 toxicities attributable to the study drugs are included in the analysis, apart from those starting after strategy failure.
  The TWiST state is defined as DDC time minus time with toxicities.
  The duration of the relapse or REL state is defined as OS time minus DDC time, or the period of time from progression to death. Patients alive at the end of the study are censored for the OS endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy NEUZILLET, MD, Principal Investigator — Institut Curie site de Saint Cloud
Locations (28):
- France (28):
  - Clinique de l'Europe, Amiens
  - Hôpital Sud CHU Amiens, Amiens
  - CH Beauvais, Beauvais
  - CHRU Jean Minjoz, Besançon
  - Clinique Tivoli Ducos, Bordeaux
  - CHU Morvan, Brest
  - GHPSO Site de Creil, Creil
  - Hôpital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHU Dijon, Dijon
  - CHRU Lille, Lille
  - centre Léon Bérard, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital la Croix Rousse, Lyon
  - Hôpital Lyon Sud Hospices Civils de Lyon, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Européen, Marseille
  - Institut Paoli Calmette, Marseille
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - CHU Robert Debré, Reims
  - Institut Curie, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Clinique Pasteur, Toulouse
  - Hôpital TROUSSEAU, Tours
  - Insitut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No